CLINICAL TRIAL: NCT07153692
Title: Clinical Efficacy and Mechanism of tDCS for Dysphagia in Patients With Parkinson's Disease
Brief Title: Clinical Efficacy and Mechanism of tDCS for Dysphagia in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Ping (Other)
Responsible Party: Sponsor-Investigator, Wang Ping, senior therapist, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: （2024）lunshenyan（1309）
Record Dates: First submitted 2025-08-05; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease and Parkinsonism; Dysphagia
Keywords: Parkinson's disease; Atypical Parkinsonian Syndromes; dysphagia; tDCS; VFSS
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Deglutition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS group (Experimental): tDCS Treatment Protocol The anode of the electrode pad will be placed on the swallowing sensorimotor cortex (S1/M1). The cathode will be placed on the contralateral supraorbital margin. The S1/M1 areas of the left and right hemispheres will be stimulated alternately, with a current intensity of 1.6mA. The treatment will be given once daily, 20 minutes per session, 5 times a week, for 2 consecutive weeks, totaling 10 sessions (5 sessions for each hemisphere).
  Conventional Dysphagia Treatment
  1. Training for perioral muscles, tongue sensory and motor functions, including ice cotton swab stimulation, gustatory stimulation, tongue muscle movement training, etc.;
  2. Airway protection training, including Mendelsohn maneuver, supraglottic swallow training, etc.;
  Interventions: Device: tDCS; Behavioral: Conventional Dysphagia Treatment
- sham tDCS group (Sham Comparator): Sham tDCS Treatment Protocol The electrode positions and treatment frequency of sham tDCS will be the same as those of real tDCS. The current is 0.05 mA. The treatment will be given once daily, 20 minutes per session, 5 times a week, for 2 consecutive weeks, totaling 10 sessions (5 sessions for each hemisphere).
  Conventional Dysphagia Treatment
  1. Training for perioral muscles, tongue sensory and motor functions, including ice cotton swab stimulation, gustatory stimulation, tongue muscle movement training, etc.;
  2. Airway protection training, including Mendelsohn maneuver, supraglottic swallow training, etc.;
  Interventions: Behavioral: Conventional Dysphagia Treatment; Device: sham tDCS

INTERVENTIONS:
Device: tDCS — The IS200 intelligent electrical stimulator, manufactured in Chengdu, Sichuan, will be used. The electrode pads are 4cm × 6cm in size. The anode of the electrode pad will be placed on the swallowing sensorimotor cortex (S1/M1). The specific positioning will follow the international 10-20 electroencephalographic system: the left S1/M1 area is located at the midpoint of the line connecting C3 and T3 in the left hemisphere; the right S1/M1 area is located at the midpoint of the line connecting C4 and T4 in the right hemisphere. The cathode will be placed on the contralateral supraorbital margin. The S1/M1 areas of the left and right hemispheres will be stimulated alternately, with a current intensity of 1.6mA. The treatment will be given once daily, 20 minutes per session, 5 times a week, for 2 consecutive weeks, totaling 10 sessions (5 sessions for each hemisphere).
  Arms: real tDCS group
Behavioral: Conventional Dysphagia Treatment — 1. Training for perioral muscles, tongue sensory and motor functions, including ice cotton swab stimulation, gustatory stimulation, tongue muscle movement training, etc.;
  2. Airway protection training, including Mendelsohn maneuver, supraglottic swallow training, etc.;
Device: sham tDCS — According to previous literature, the electrode positions and treatment frequency of sham tDCS will be the same as those of real tDCS. The current will be adjusted to 0.05mA.
  Arms: sham tDCS group

SUMMARY:
This study aims to verify transcranial direct current stimulation(tDCS) efficacy for Parkinson's disease (PD)-related dysphagia and its mechanism. Subjects are randomly split into two groups: control (sham tDCS + conventional dysphagia treatment) and experimental (real tDCS + conventional treatment).

Assessments will be conducted at baseline, after the completion of intervention, and at the 3-month follow-up. Swallowing function will be evaluated via gold-standard videofluoroscopic swallowing study (VFSS) and scales. Resting-state functional magnetic resonance imaging (rs-fMRI) or functional near-infrared spectroscopy (fNIRS) will be measures for tracking changes in abnormal brain regions/networks.

Correlations between swallowing recovery and brain function changes, plus group imaging differences, will reveal tDCS's neurophysiological mechanism.

DETAILED DESCRIPTION:
This study aims to verify the efficacy of tDCS in treating dysphagia in PD and explore its mechanism. Subjects are randomly divided into two groups: the control group receives sham tDCS as well as the conventional dysphagia treatment, while the experimental group undergoes real tDCS combined with conventional dysphagia treatment.

All subjects will be evaluated before treatment, after treatment, and 3 months later (follow-up). Swallowing function in both groups will be assessed using the gold standard VFSS and swallowing scales. Additionally, techniques including amplitude of low frequency fluctuation (ALFF) and functional connectivity (FC) in rs-fMRI or fNIRS will be used to observe changes in abnormal brain regions and brain network connectivity before and after treatment in both groups.

This study will also explore the correlation between swallowing function recovery and the alteration of brain function, compare the imaging differences between the two groups, and thereby reveal the neurophysiological mechanism underlying tDCS in the treatment of PD-related dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Chinese Diagnostic Criteria for Parkinson's Disease (2016) or MDS Diagnostic Criteria for Multiple System Atrophy or Progressive Supranuclear Palsy;
* VFSS examination indicates dysphagia;
* Mini-Mental State Examination (MMSE) score >23;
* Willing to cooperate with the study and sign the informed consent form;

Exclusion Criteria:

* Comorbid with other diseases that cause dysphagia;
* Comorbid with pneumonia, or severe cardiac/renal insufficiency;
* Having metal implants in the body
* With cognitive impairment or inability to cooperate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Rosenbek Penetration-Aspiration Scale (PAS): | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  Scored 1-8, with higher scores indicating poorer swallowing safety.
  1. Level 1: The bolus does not enter the airway; it remains entirely within the oral cavity or pharynx and is propelled normally.
  2. Level 2: The bolus enters the supraglottic area (e.g., vallecula) but does not touch the vocal cords, and is completely cleared (e.g., via swallowing or coughing).
  3. Level 3: The bolus enters the supraglottic area without touching the vocal cords, but residue remains (not fully cleared).
  4. Level 4: The bolus touches the vocal cords but does not enter the subglottic airway, and is completely cleared.
  5. Level 5: The bolus touches the vocal cords without entering the subglottic airway, but residue remains.
  6. Level 6: The bolus enters the subglottic airway (into the trachea) but is completely cleared by the patient (e.g., via coughing).
  7. Level 7: The bolus enters the subglottic airway; the patient exhibits protective responses (e.g., coughing) but cannot fully clear it, leaving
Videofluoroscopic Dysphagia Scale (VDS) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  14 items in total, including 7 items for oral-phase swallowing function and 7 for pharyngeal-phase function, used to assess overall swallowing function;
oral residue | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  Post-swallow residue was scored 0-3, with higher scores indicating more food residue and lower swallowing efficiency
Amplitude of Low Frequency Fluctuation (ALFF) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  ALFF focuses on the low-frequency components of these HbO/HbR time series. It is defined as the average amplitude of hemodynamic signal fluctuations within a specific low-frequency range (typically 0.01-0.1 Hz, though the exact band may vary by study). This range is chosen because it captures slow, spontaneous oscillations in cerebral blood flow and oxygenation, which are hypothesized to reflect synchronized neural activity across brain regions (e.g., default mode network, sensorimotor networks).
  Mathematically, ALFF quantifies the "strength" of these low-frequency oscillations: a higher ALFF value indicates more prominent or intense fluctuations in the target frequency band, suggesting greater spontaneous hemodynamic (and thus neural) activity in that brain region.
Functional Connectivity (FC) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  Functional Connectivity (FC) refers to the statistical association or synchronization between spontaneous hemodynamic signals from different cortical regions, reflecting the coordinated activity of spatially distinct brain areas. It quantifies how closely the neural activity (inferred from blood oxygenation changes) in one brain region correlates with that in another, providing insights into the integration of brain networks.
vellaculae residue | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  The residue amount was rated on a scale from 0 to 3: 0 indicates that no residue was visible, 1 indicates mild residue(the level of contrasted material constituted less than 25% of the height of the structure), 2 indicates moderate residue (the level of contrasted material constituted between 25 and 50%of the height of the structure), and 3 indicates severe residue(the level was higher than 50% of the height of the structure).
pyriform sinuses residue | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  The residue amount was rated on a scale from 0 to 3: 0 indicates that no residue was visible, 1 indicates mild residue(the level of contrasted material constituted less than 25% of the height of the structure), 2 indicates moderate residue (the level of contrasted material constituted between 25 and 50%of the height of the structure), and 3 indicates severe residue(the level was higher than 50% of the height of the structure).

SECONDARY OUTCOMES:
temporal indicators | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  TT, PTT, LVCrt, and so on.
spatial indicators | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  hyoid bone advancement, hyoid bone elevation, PCR
Swallowing Disorder Questionnaire (SDQ) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  A swallowing function screening scale with 15 items, scored up to 44.5; higher scores indicate more severe dysphagia.
Functional Oral Intake Scale (FOIS) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  7 levels in total, with Level 1 indicating the most severe feeding impairment and Level 7 indicating normal function.

OTHER OUTCOMES:
Unified Parkinson's Disease Rating Scale-III (UPDRS-III) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  14 items, scored up to 56; higher scores indicate more severe motor dysfunction.
Swallowing Quality of Life Questionnaire (SWAL-QOL) | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  The SWAL-QOL is a patient-reported outcome tool designed to assess the impact of oropharyngeal dysphagia on health-related quality of life. It Comprises 44 items. it evaluates both subjective experiences (e.g., psychological burden) and clinical symptoms (e.g., choking, food sticking) through self-reported responses.
Non-Motor Symptoms Scale (NMSS) for Parkinson's Disease | at baseline, after the completion of 10 days of intervention, at the 3-month follow-up
  30 items, scored up to 210; higher scores indicate more severe non-motor symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Wang, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan includes making the statistical results of the data publicly available to other researchers.

REFERENCES:
- [Result] Ding X, Gao J, Xie C, Xiong B, Wu S, Cen Z, Lou Y, Lou D, Xie F, Luo W. Prevalence and clinical correlation of dysphagia in Parkinson disease: a study on Chinese patients. Eur J Clin Nutr. 2018 Jan;72(1):82-86. doi: 10.1038/ejcn.2017.100. Epub 2017 Jul 12. PMID 28699630
- [Result] Henry KA, Singh R, Zhang N, Lyons MK, McNett K, Neal MT, Mehta SH. Effect of STN/GPi DBS on swallowing function in Parkinson's disease as assessed by Video fluoroscopy: A retrospective study. Parkinsonism Relat Disord. 2022 Oct;103:136-140. doi: 10.1016/j.parkreldis.2022.08.017. Epub 2022 Sep 11. PMID 36115199
- [Result] Wang P, Wang B, Chen X, Xiong B, Xie F, Wu S, Tang Y, Chen S, Ding X, Liu P, Luo W. Six-Year Follow-Up of Dysphagia in Patients with Parkinson's Disease. Dysphagia. 2022 Oct;37(5):1271-1278. doi: 10.1007/s00455-021-10387-0. Epub 2021 Nov 26. PMID 34826007
- [Result] Gandhi P, Steele CM. Effectiveness of Interventions for Dysphagia in Parkinson Disease: A Systematic Review. Am J Speech Lang Pathol. 2022 Jan 18;31(1):463-485. doi: 10.1044/2021_AJSLP-21-00145. Epub 2021 Dec 10. PMID 34890260
- [Result] Dashtelei AA, Nitsche MA, Salehinejad MA, Habibi AH, Bakhtyiari J, Khatoonabadi AR. Adjunctive transcranial direct current stimulation to improve swallowing functions in Parkinson's disease. EXCLI J. 2024 Jan 18;23:95-107. doi: 10.17179/excli2023-6496. eCollection 2024. PMID 38487086